CLINICAL TRIAL: NCT05566691
Title: Strategies for Coping With Negative Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022B0242
Record Dates: First submitted 2022-09-02; First posted 2022-10-04 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Depressive Symptoms; Anxiety; Negative Thinking
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Positive thinking (Active Comparator): Videos will describe negative automatic thoughts and then describe positive thinking, its benefits, and how to use it to cope with negative thoughts. A worksheet will then walk participants through applying the strategy to a recent negative thought of their own. Daily surveys will involve a shortened version of this worksheet.
  Interventions: Other: Positive thinking
- Positive thinking plus mood induction (Active Comparator): The same videos will be used to describe negative automatic thoughts and then describe positive thinking, its benefits, and how to use it to cope with negative thoughts. Participants will then undergo a positive mood induction in which they are asked to recall a pleasant memory and try to re-experience those feelings. A worksheet will then walk participants through applying the strategy to a recent negative thought of their own. Daily surveys will involve the same mood induction and a shortened version of this worksheet.
  Interventions: Other: Positive thinking + Mood induction
- Thought reevaluation (Active Comparator): Videos will describe negative automatic thoughts and then describe reevaluating thoughts, its benefits, and how to use it to cope with negative thoughts. A worksheet will then walk participants through applying the strategy to a recent negative thought of their own. Daily surveys will involve a shortened version of this worksheet.
  Interventions: Other: Thought reevaluation
- Thought reevaluation plus mood induction (Active Comparator): The same videos will be used to describe negative automatic thoughts and then describe reevaluating thoughts, its benefits, and how to use it to cope with negative thoughts. Participants will then undergo a positive mood induction in which they are asked to recall a pleasant memory and try to re-experience those feelings. A worksheet will then walk participants through applying the strategy to a recent negative thought of their own. Daily surveys will involve the same mood induction and a shortened version of this worksheet.
  Interventions: Other: Thought reevaluation + Mood induction

INTERVENTIONS:
Other: Positive thinking — Participants will be provided with information about how to cope with negative thoughts using positive thinking and asked to complete a worksheet walking them through the steps of positively reevaluating negative thoughts.
  Arms: Positive thinking
Other: Positive thinking + Mood induction — Participants will be provided with information about how to cope with negative thoughts using positive thinking and asked to complete a worksheet walking them through the steps of positively reevaluating negative thoughts. They will be assigned to a positive mood induction before completion of the worksheet.
  Arms: Positive thinking plus mood induction
Other: Thought reevaluation — Participants will be provided with information about how to cope with negative thoughts using thought reevaluation and asked to complete a worksheet walking them through the steps of reevaluating negative thoughts.
  Arms: Thought reevaluation
Other: Thought reevaluation + Mood induction — Participants will be provided with information about how to cope with negative thoughts using thought reevaluation and asked to complete a worksheet walking them through the steps of reevaluating negative thoughts. They will be assigned to a positive mood induction before completion of the worksheet.
  Arms: Thought reevaluation plus mood induction

SUMMARY:
The primary objective of this study is to assess the impact of two strategies for coping with negative automatic thoughts (positive thinking and cognitive restructuring) on one's belief in negative thoughts and one's affect. Another main objective is to assess whether participating in a positive mood induction (versus no mood induction) prior to using one of the two coping strategies impacts belief in negative thoughts and affect. We will also explore the interaction between strategy condition and mood induction condition. As secondary outcomes, we will evaluate whether there are changes in positive thinking skills and cognitive restructuring skills and depressive symptoms after one week of using the strategy.

DETAILED DESCRIPTION:
Participants will be randomized to learn about positive thinking or cognitive restructuring, which will involve watching brief videos, being presented with examples of how one might apply the strategy when experiencing negative thoughts, and practicing with a personal example using a worksheet. Participants will also be randomized to positive mood induction, which is comprised of an autobiographical recall exercise in which participants are asked to recall a pleasant memory before filling out the worksheet. Participants will be asked to use the strategy and complete a worksheet online once per day for six days. Participants will respond to questionnaires at baseline and after 6 days of strategy use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older.

Exclusion Criteria:

* A level of visual impairment that would prevent them from being able to answer questions on an electronic screen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule | Assessed at baseline, each day for 6 days, and one week post-baseline.
  The PANAS is a 20-item self report scale that measures positive affect (10 items) and negative affect (10 items). Each item is rated on a Likert scale from 1 to 5, with higher scores indicating a higher endorsement of each affective descriptor.
Change in belief in negative thought | Assessed at baseline, each day for 6 days, and one week post-baseline.
  Participants will be asked how much they believed in a negative thought (0-100%) they recently experienced before completing a worksheet. After using a positive thinking or cognitive restructuring worksheet, participants will rate how much they currently believe their initial negative thought.
Change in mood | Assessed at baseline, each day for 6 days, and one week post-baseline.
  Participants will be asked to rate their mood on a scale of 0 (very negative) to 100 (very positive) before and after the positive mood induction.

SECONDARY OUTCOMES:
Change in positive thinking and cognitive restructuring skills | Assessed at baseline and one week post-baseline.
  Cognitive restructuring skills will be assessed by the Competencies of Cognitive Therapy Scale-10, which is a 10-item self-report measure assessing the use of cognitive strategies to cope with negative mood. Positive thinking skills will be measured by the 10-item Positive Thinking Skills Scale, which assesses the use of positive thinking strategies to cope with negative mood.
Change in Quick Inventory of Depressive Symptoms Self-Report | Assessed at baseline and one week post-baseline.
  The QIDS-SR is a 16-item self-report measure of depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater depressive symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05566691/ICF_000.pdf